CLINICAL TRIAL: NCT06305221
Title: Effect of Opioid-free Analgesia and Anesthesia on the Quality of Postoperative Recovery and Nausea Vomit in Patients Receiving Laparoscopic Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bijia Song, principal investigator, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: opioid-free analgesia
Record Dates: First submitted 2024-03-03; First posted 2024-03-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Opioid-Free Anesthesia; Laparoscopic Sleeve Gastrectomy; Postoperative Vomiting; Postoperative Recovery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Esketamine; Dexmedetomidine; Sufentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free group (Experimental)
  Interventions: Drug: Opioid-free Analgesics (esketamine, dexmedetomidine)
- Opioid group (Active Comparator)
  Interventions: Drug: Opioid Anesthetics (sufentanil and remifentanil)

INTERVENTIONS:
Drug: Opioid-free Analgesics (esketamine, dexmedetomidine) — opioid free group: After infusion of a loading dose of dexmedetomidine, intravenous midazolam 2mg, propofol 2mg kg-1, esketamine 0.5 mg kg-1, rocuronium 0.6-1mg kg-1, and 3min after endotracheal intubation. Intravenous continuous infusion of propofol, esketamine and dexmedetomidine hydrochloride mixture (esketamine 50mg + dexmedetomidine hydrochloride 150 ug + 0.9% saline 50ml in the same 50ml syringe) 0.1ml kg-1 h-1-0.2 ml kg-1 h-1 (equivalent to esketamine 0.1-0.2mg kg-1 h-1; Dexmedetomidine hydrochloride 0.3-0.6 μ g kg-1 h-1) maintains a BIS value between 40-60, 10-20mg / time was added as appropriate.
  Arms: Opioid-free group
Drug: Opioid Anesthetics (sufentanil and remifentanil) — Intravenous midazolam 2mg, propofol 2mg kg-1, sufentanyl 0.3-0.5 μ g kg-1, rocuronium 0.6-1mg kg-1,3min before endotracheal intubation. After successful endotracheal intubation, continuous intravenous infusion of propofol and remifentanil was started to maintain BIS values between 40-60, and rocuronium 10-20mg / time as appropriate. After the start of surgery, 10-20 μ g of sufentanil was added according to blood pressure and heart rate. At the end of the operation, 5mg and 50mg were injected before the end of the operation, and propofol and remifentanil were stopped at the end of the operation
  Arms: Opioid group

SUMMARY:
The purpose of the intraoperative use of opioids is to reduce the amount of sedative medication and to ensure effective analgesia. But pain is an unpleasant sensory and emotional experience (a cognitive perception) that cannot occur with sufficient depth of anesthesia (even without opioids). So a more reasonable explanation for analgesia should be anti-nociception and the resulting inhibition of the response to surgical stress. Since multiple mediators are involved in nociceptive pathways, antinociception can also be acquired through multiple mechanisms. However, there is no single ideal harm drug to replace opioids, which often requires two or more drugs to meet clinical needs. While regional block attenuates the stress response to surgery and sympathetic activation because of afferents to block nociceptive stimuli, and has an important role in the implementation of OFA. Combined with the clinical characteristics of the LSG, investigators developed the transverse abdominis fascia block (transversus abdominis plane TAP) in combination with esketamine (esketamine), dexmedetomidine (dexmedetomidine, DEX) of opioid-free anesthesia (opioid free anesthesia, OFA) and the analgesic regimen (TEDOFA), Reduce patient pain scores, nausea and vomiting after LSG based on perfect analgesia and adequate anti-sympathetic response, As well as the other complications, Promote the accelerated postoperative recovery of patients undergoing LSG, And reduce the incidence and severity of postoperative chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic sleeve gastrectomy

  * ASAA I or grade;

    * volunteered in this trial and signed informed consent; ④ age 18-65 years; ⑤ BMI> 30kg / m2.

Exclusion Criteria:

* chronic pain;
* severe liver dysfunction (total bilirubin 2 mg dl-1);
* severe renal dysfunction (glomerular filtration rate 60ml min-1 1.73m-2);
* pregnancy or lactation;
* preoperative heart rate <50 beats / min, sick sinus syndrome, severe heart block; -dementia or significant neurological disorders (such as stroke, epilepsy, intracranial tumors, PD, etc.);
* history of alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
15-item recovery quality scale score 48 hours after surgery | 48 hours after surgery
  The QoR-15 scale is a global measure of postoperative recovery, with scores ranging from 0 (extremely poor QoR) to 150 (excellent QoR). QoR-15 has become the most widely reported indicator for the evaluation of postoperative life treatment in patients. Using wherever possible QoR-15 item scores on postoperative day 3, QoR-15 with very good validity, and good reliability, responsiveness and clinical acceptability, these data suggest that QoR-15 is an excellent patient-centered measure of postoperative QoR. Patient Acceptable symptom status describes the lowest absolute score considered by the patient to represent a healthy or good status health scale. A QoR-15 score of 118 or more indicates a good postoperative recovery
15-item recovery quality scale score 24 hours before surgery | 24 hours before surgery
  The QoR-15 scale is a global measure of postoperative recovery, with scores ranging from 0 (extremely poor QoR) to 150 (excellent QoR). QoR-15 has become the most widely reported indicator for the evaluation of postoperative life treatment in patients. Using wherever possible QoR-15 item scores on postoperative day 3, QoR-15 with very good validity, and good reliability, responsiveness and clinical acceptability, these data suggest that QoR-15 is an excellent patient-centered measure of postoperative QoR. Patient Acceptable symptom status describes the lowest absolute score considered by the patient to represent a healthy or good status health scale. A QoR-15 score of 118 or more indicates a good postoperative recovery
15-item recovery quality scale score 24 hours after surgery | 24 hours after surgery
  The QoR-15 scale is a global measure of postoperative recovery, with scores ranging from 0 (extremely poor QoR) to 150 (excellent QoR). QoR-15 has become the most widely reported indicator for the evaluation of postoperative life treatment in patients. Using wherever possible QoR-15 item scores on postoperative day 3, QoR-15 with very good validity, and good reliability, responsiveness and clinical acceptability, these data suggest that QoR-15 is an excellent patient-centered measure of postoperative QoR. Patient Acceptable symptom status describes the lowest absolute score considered by the patient to represent a healthy or good status health scale. A QoR-15 score of 118 or more indicates a good postoperative recovery

SECONDARY OUTCOMES:
Dosage of postoperative analgesics | 48 hours after surgery
  record dosage of postoperative analgesics
Duration of until postoperative PACU Aldrete score> 9 points | up to 30 min after surgery at postoperative recovery room
  Anesthesia recovery was defined by Aldrete's recovery score (RS, 0-10), assessed following postanesthesia care unit (PACU) arrival, with RS ≥9 considered discharge eligible
anesthesia-related complication | 24 hours after surgery
  record anesthesia-related complication
time to first exhaust gas after surgery | 24 hours after surgery
time of first postoperative mobilization | 24 hours after surgery
Overall benefit of analgesic score satisfaction in pain treatment | 6, 24, 48 hours after surgery
  To calculate the OBAS score, compute the sum of scores in items 1-6 and add '4-score in item 7'. Note that a low score indicates high benefit. test overall benefit of analgesic score satisfaction in pain treatment at 6, 24, 48 hours after surgery
Acute pain numeric rating scale score | 6, 24, 48 hours after surgery
  The pain 0-10 classification is the numerical classification (NRS) of subjective assessment, with 0 painless pain, 1-3 mild pain, 4-6 moderate pain, 7-9 severe pain, and 10 severe pain. test acute pain numeric rating scale score at 6, 24, 48 hours after surgery
Rhodes Index of Nausea, Vomiting, and Retching | one night before surgery
  Rhodes Index of Nausea, Vomiting, and Retching, an 8-item questionnaire, to measure the incidence and severity of nausea, vomiting, and retching At each timepoint, a total Rhodes score was calculated from the sum of the 8 RINVR questions. Total Rhodes scores were compared at 6 different timepoints as well as overall across all 6 time points. record Nausea and vomiting, the Rhodes index score
Rhodes Index of Nausea, Vomiting, and Retching | 6, 24, 48 hours after surgery
  Rhodes Index of Nausea, Vomiting, and Retching , an 8-item questionnaire, to measure the incidence and severity of nausea, vomiting, and retching At each timepoint, a total Rhodes score was calculated from the sum of the 8 RINVR questions. Total Rhodes scores were compared at 6 different timepoints as well as overall across all 6 time points. record Nausea and vomiting, the Rhodes index score. record Nausea and vomiting, the Rhodes index score

CONTACTS AND LOCATIONS:
Locations (1):
- bijia Song, Beijing, China